CLINICAL TRIAL: NCT05619120
Title: Potential of Late Na Current Blocker Mexilate on Giant T-wave Electrical Alternans and Subsequent Ventricular Arrhythmias: a Multicenter, Randomized, Prospective Study
Brief Title: The Effect of Late Na Current Blocker Mexiletine on Giant T-wave Electrical Alternans(STOP-TWA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2021CRF-001
Record Dates: First submitted 2019-11-24; First posted 2022-11-16 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Giant T-wave Electrical Alternans
MeSH Terms: interventions — Mexiletine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giant T-wave electrical alternans conventional plus mexiletine therapy (Experimental): It is proposed that patients presenting with giant TWA-triggered VT/VF patients to be randomized to conventional treatment and conventional plus mexiletine treatment, respectively.
  Interventions: Drug: Mexiletine; Other: Conventional therapy
- Giant T-wave electrical alternans conventional therapy (Active Comparator): Conventional treatment in the control group according to the guidelines for the management of ventricular arrhythmias (2017 AHA/ACC/HRS)
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Drug: Mexiletine — Mexiletine (150mg, bid, po) is given to patients who have been divided into Mexiletine group.
  Arms: Giant T-wave electrical alternans conventional plus mexiletine therapy
Other: Conventional therapy — Treatment according to the guidelines for the management of ventricular arrhythmias (2017 AHA/ACC/HRS)

SUMMARY:
The electrocardiogram is one of the most basic tests for cardiovascular disease. T wave alternans (TWA), which reflects abnormal ventricular repolarization, can easily trigger ventricular tachycardia (VT) and ventricular fibrillation (VF), which are important warning clues for sudden cardiac death (SCD). The late sodium current (INaL) is an important component of the frequency-dependent regulation of cardiac repolarization, and various causes of delayed repolarization can increase INaL. Our study on long QT syndrome (LQTS) found that INaL abnormalities can lead to abnormal myocardial repolarization, producing a giant TWA that triggers VT and VF. VT and VF, and INaL inhibition by the INaL blocker mexilate can terminate this process. This suggests that pharmacological blockade of INaL may be a potential target for the prevention of SCD by ameliorating the different causes of giant TWA and its triggering ventricular arrhythmic events. In this study, we propose to randomize patients with VT/VF triggered by giant TWA to conventional treatment and conventional treatment adds mexiletine treatment to compare the effects of the two treatment regimens on giant TWA and its triggered nonsustained VT, sustained VT, and VF; at the same time, we will compare the effects of mexiletine on giant TWA and its triggered ventricular arrhythmias of various etiologies by intra-group control before and after treatment. The safety and efficacy of the treatment of TWA and its triggered ventricular arrhythmias are compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of macroscopic TWA

Exclusion Criteria:

* The patients who do not agree to participate in the study,
* Patients with acute coronary syndrome or with progressive myocardial ischemia according to clinical manifestations, electrocardiogram or myocardial biochemical markers;
* Those who have used other class I antiarrhythmic drugs or who are contraindicated by mexiletine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the occurrence of macroscopic TWA | at administration,1，2，3，4，5，6，7 days after administration.
  Macroscopic TWA occurring on conventional ECG (12-lead ECG, telemetry ECG, or holter ECG) with visually identifiable TWA Diagnosis confirmed by at least 3 leading ECG specialists. The data is obtained from the medical records.

SECONDARY OUTCOMES:
Length of hospital stay | About 7 days after administration.
  Comparison between two treatment groups due to the effect of ventricular arrhythmia episodes on the duration of hospitalization ( days) in patients. The data is obtained from the medical records.
Change in the number of refractory cases | At administration,1，2，3，4，5，6，7 days after administration.
  The number of cases in the group requiring ICD for ventricular arrhythmia episodes. The data is obtained from the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital of Xi'an Jiaotong University, China
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No